CLINICAL TRIAL: NCT01236677
Title: The Establishment and Improvement of Community Acquired Pneumonia Monitoring and Disposal Network in Beijing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Chen Wang, Capital Medical University Affiliated Beijing Chaoyang Hospital
Other Study IDs: xfcrb123456
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-08

CONDITIONS: Community Acquired Pneumonia
Keywords: Pathogen
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sputum,serum,and throat swabs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Community acquired pneumonia,age≥14 ys: Patients with community acquired pneumonia,age≥14 ys and less than one week after the onset of symptoms, without pregnancy,breast-feeding,HIV infection,recent 90-day hospitalized history and in nursing homes or rehabilitation hospitals

SUMMARY:
In the 21st century, threats to human health of new respiratory infectious diseases increased.

The project aim is to establish pneumonia pathogens network in Beijing and understand the pathogen spectrum distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed community acquired pneumonia
2. Age≥14 ys
3. New appear of cough or cough become severe
4. New infiltration showed by chest radiology(x-ray or CT)
5. Fever T>37.8o C or <35.6o C
6. White blood cell>10,000/mm3 , left shift or leukopenia<4000/ul）

Exclusion Criteria:

1. Pregnancy or breast-feeding
2. Over one week after the onset of symptoms
3. HIV infection
4. Recent 90-day hospitalized history(length of stay greater than 2 days)
5. Live in nursing homes or rehabilitation hospitals

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Confirmed community acquired pneumonia
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of all symptoms (defined as the period from start of study-drug to relief of fever) | one year

SECONDARY OUTCOMES:
If duration of symptoms long, follow-up 30 days. | one year
In case of early termination:death;diagnosed tuberculosis;diagnosed lung cancer and HIV infection | one year

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Doctor, Study Chair — Capital Medical University affiliated Beijing Chaoyang Hospital, Beijing Respiratory Medicine Insititute
Locations (1):
- Capital Medical University affiliated Beijing Chaoyang Hospital, Beijing Respiratory Medicine Insititute, Beijing, Beijing Municipality, China